CLINICAL TRIAL: NCT05527951
Title: Enhanced Measurement-Based Care Effectiveness for Depression (EMBED) Study:A Cluster Randomized Controlled Trial of Enhanced Versus Standard Measurement-Based Care Implementation for Depression
Brief Title: Enhanced Measurement-Based Care Effectiveness for Depression (EMBED) Study
Acronym: EMBED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: University of British Columbia (Other); University of Toronto (Other); University of Melbourne (Other); Boston University (Other); University of California (Other); University of Alberta (Other); Shanghai CDC for Mental Health (Unknown); Institute of Population Research, Peking University (Unknown); University of Michigan (Other); Queen's University (Other); Hongkou Mental Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-77
Record Dates: First submitted 2022-08-11; First posted 2022-09-06 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-07

CONDITIONS: Major Depressive Disorder
Keywords: measurement-based care; scales; assessment; depression; randomized; cluster trial; implementation; mobile health; WeChat; clinical trial; mixed methods; China
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: The study protocol involves a 2-arm cluster RCT of enhanced versus standard measurement-based care implementation for depression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced MBC Implementation(eMBC) (Experimental): The eMBC implementation arm use our WeChat Easy to Recover from Depression Mini-Program, which consists of mood tracking and lay-coached self-management.
  Interventions: Other: eMBC
- Standard MBC Implementation (Active Comparator): The standard MBC implementation arm use paper and pencil questionnaires.
  Interventions: Other: standard MBC

INTERVENTIONS:
Other: eMBC — The experimental group will implement eMBC with our WeChat Easy to Recover from Depression Mini-Program, which consists of mood tracking and lay-coached self-management.
  Arms: Enhanced MBC Implementation(eMBC)
Other: standard MBC — The control intervention group will implement standard MBC using paper and pencil questionnaires.
  Arms: Standard MBC Implementation

SUMMARY:
Measurement-based care (MBC) is an evidence-based practice that incorporates routine outcome assessment using validated rating scales to guide collaborative clinical decision-making. Although MBC results in improved outcomes for patients with major depressive disorder (MDD), there are barriers to its broad implementation in clinical settings. The use of "enhanced" MBC (eMBC), with mobile apps that allow patients to track outcomes and engage in self-management via WeChat, may address some of these barriers. The investigators hypothesize that implementation with eMBC using WeChat will be superior to standard MBC implementation using paper-pencil assessments at the clinic, for both implementation and clinical outcomes.

DETAILED DESCRIPTION:
The investigators present a trial protocol for a 2-arm cluster randomized controlled trial (RCT) with a hybrid implementation-effectiveness design comparing standard MBC implementation versus eMBC implementation with 6-month follow up in 12 mental health centers in Shanghai, China. The eMBC implementation uses a WeChat mini-program that includes outcome tracking using brief questionnaires and self-management lessons supplemented with support by a lay coach via WeChat.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-65 years;
2. Participants were diagnosed of unipolar depressive disorder by the treating physician based on accepted diagnostic criteria (e.g., CCMD-3, DSM-IV, DSM-5, ICD-10);
3. Participants are expected to have a smartphone device available and be proficient in using a smartphone;
4. Participants should have a junior high school education or above, have sufficient audio-visual skills, be able to fully understand the research content and have the legal ability to sign informed consent.

Exclusion Criteria:

1. Presence of obvious violent aggressive behavior or tendencies;
2. Participants who are unstable during onset episodes and cannot cooperate in completing the study content;
3. Serious suicidal tendencies;
4. Inability to carry out effective verbal communication;
5. No smartphone;
6. Other circumstances that prevented cooperation or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | up to 6 months
  To evaluate the severity of depressive symptoms by patients. Remission: total score ≤ 4.
Proportion of patients with a Patient Health Questionnaire-9 (PHQ-9) score | up to 6 months
  Proportion of patients with a PHQ-9 score entered in the clinical record.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9(PHQ-9) change scores | up to 6 months
  The changes in PHQ-9 scores and depression categories were determined by subtracting the final PHQ-9 score from the initial PHQ-9 score. Therefore, a negative change in PHQ-9 represents a lessening of depression symptoms while a positive change in PHQ-9 represents an increase in depression symptoms.
The Sheehan disability scale (SDS) | up to 6 months
  To evaluate the functional impairment, including work/study, daily life and family responsibility. The score of each subscale ranged from 0 to 10 which means from no impairment to loss of function.
Quality of Life scale (QOL-6) | up to 6 months
  To evaluate the quality of life in patients with MDD. The higher the total score, the better the quality of life.
EuroQoL 5 Dimensions (EQ-5D) | up to 6 months
  To evaluate the quality of life in patients with MDD. The higher the total score, the better the quality of life.
Health economic assessment (HEA) | up to 6 months
  To evaluate the health services utilization. Economic outcomes will include health service utilization data (both mental health- and non-mental health-related) from the HEA and from available EMR/chart records, including health provider encounters, emergency room visits, hospitalizations, diagnostic tests, and prescriptions.
Patient Adherence Questionnaire(PAQ) | up to 6 months
  To evaluate the medication adherence.The PAQ is a two item measure, with the first question assessing level of adherence (quantified as number of days in the past week in which medication was not taken) and item 2 assesses reasons for non-adherence.
Scale To Assess Therapeutic Relationships in Community Mental Health Care (STAR-P) | up to 6 months
  To assess the therapeutic relationship between patients and clinicians in community mental health care settings.It contains 12 items and each item is rated on a 5-point Likert scale, with answers ranging from 0 to 4.
Proportion of patients who accessed the WeChat Easy to Recover from Depression Mini-Program at least once | up to 6 months
  Proportion of patients who accessed the WeChat Easy to Recover from Depression Mini-Program at least once.
Proportion of patients who completed at least 4 of 6 lessons in Come Back mini-program | up to 6 months
  Proportion of patients who completed at least 4 of 6 lessons in the Come Back mini-program.Come Back mini-program is a part of the WeChat Easy to Recover from Depression Mini-Program,which consists of 6 weekly lessons based on cognitive-behavioural therapy (CBT) principles.
System Usability Scale | up to 6 months
  To evaluate patient satisfaction by qualitative interviews.Participants are asked to score 10 items with one of five responses that range from Strongly Agree to Strongly disagree.
Evidence Based Practice Attitude Scale (EBPAS) | up to 6 months
  To evaluate clinician satisfaction by qualitative interviews.Participants are asked to score 15 items with one of five responses that range from Not at All to To a Very Great Extent.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center(SMHC)
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam RW, Michalak EE, Murphy JK, Colquhoun H, Ng C, Culpepper L, Dewa CS, Greenshaw AJ, He Y, Kennedy SH, Li X, Liu J, Liu T, Parikh S, Soares CN, Wang Z, Xu Y, Chen J. Standard Versus Enhanced Measurement-Based Care Effectiveness for Depression (EMBED): Protocol for a Cluster Randomized Implementation-Effectiveness Trial. Cureus. 2025 Aug 18;17(8):e90395. doi: 10.7759/cureus.90395. eCollection 2025 Aug. PMID 40970017